CLINICAL TRIAL: NCT03077919
Title: A Randomized, Sham-procedure-controlled, Blinded Study to Evaluate the Effectiveness and Acceptability of Right-sided Stellate Ganglion Block for Treatment of Posttraumatic Stress Disorder Symptoms
Brief Title: Effectiveness and Acceptability of Stellate Ganglion Block for Posttraumatic Stress Disorder Symptoms - Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Womack Army Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency); Landstuhl Regional Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-201
Record Dates: First submitted 2017-03-01; First posted 2017-03-13 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: PostTraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Generalized Anxiety Disorder; Depression; Distress; Alcohol Use; Pain
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Depression; Alcohol Drinking; Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be centrally randomized to 2:1 active:sham SGB and will be evaluated at Womack Army Medical Center in North Carolina, Tripler Army Medical Center in Hawaii, and Landstuhl Regional Medical Center in Germany. Randomization will be stratified by site so that each will have a 2:1 active:sham ratio. The target population includes active-duty service members and study duration is 10 weeks in the clinical effectiveness trial for which an enrollment of 240 participants is planned.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block (SGB) (Active Comparator): 7-10 mL 0.5% ropivacaine injected under ultrasound visualization ventral to right longus coli muscle (around and into the ventral fascia) and into the longus coli immediately dorsal to the presumed ventral fascia, at the level of the C6 anterior tubercle (landmarks for stellate ganglion).
  Interventions: Drug: Ropivacaine
- Sham Treatment (Sham Comparator): 1-2 mL preservative-free normal saline, injected under ultrasound visualization anterolateral to right anterior tubercle of C6.
  Interventions: Drug: Sham treatment

INTERVENTIONS:
Drug: Ropivacaine — 0.5% ropivacaine
  Other Names: Naropin
  Arms: Stellate Ganglion Block (SGB)
Drug: Sham treatment — preservative-free normal saline
  Other Names: saline
  Arms: Sham Treatment

SUMMARY:
This is a multisite, randomized, blinded, sham-procedure-controlled study to evaluate the efficacy of right-sided stellate ganglion block (SGB) on the acute symptomatology of Post traumatic Stress Disorder (PTSD), evaluated by the Clinician-Administered PTSD Scale (CAPS-5) clinical interview at pre-treatment and at 8 weeks. This entry describes the effectiveness study.The acceptability study is described in a separate entry.

DETAILED DESCRIPTION:
Study intervention will be administered at week 0 and at week 2. Injections will be performed under ultrasound visualization. The study medication will be either 7-10 mL 0.5% ropivacaine injected ventral to the right longus coli muscle (around and into the ventral fascia) and into the longus coli immediately dorsal to the presumed ventral fascia at the level of the C6 anterior tubercle (landmarks for the stellate ganglion) (active study medication) or 1-2 mL preservative free normal saline injected anterolateral to the anterior tubercle of C6 (sham procedure). The participant will not be informed which treatment he or she has received and the interaction of the participant and treating physician will be scripted as much as possible. Following the intervention, the treating physician should have no further contact with the participant except as required for participant safety.

Participants will be evaluated for posttraumatic stress disorder (PTSD) symptomatology prior to week 0 and at 8 weeks using the Diagnostic and Statistical Manual (DSM-5) Clinician-Administered PTSD Scale (CAPS-5). They will complete the PTSD Checklist for DSM-5 (PCL-5), the PTSD Checklist - Civilian Version (PCL-C), and the Mini-international Neuropsychiatric Interview (M.I.N.I.-Plus) Suicidality Items at 0, 2, 4, 6, and 8 weeks; they also will complete the M.I.N.I.-Plus items at screening. The 12 item short form survey (SF-12), generalized anxiety disorder 7-item (GAD-7), patient health questionnaire (PHQ-9), K6, Alcohol Use Disorder Identification Test (AUDIT-C/AUDIT), and a short pain scale will be completed at weeks 0, 4, and 8.

Data collected at baseline and 8 weeks will be the primary focus of data analysis. Data collected at other time points will be analyzed as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Army on active duty status
* Personal access to Internet
* Anticipated stable assignment to installation for at least 2 months
* Stable dosing for ≥3 months, if receiving psychotropic medications
* Prior to enrollment, offered PTSD treatment using A-level modality (as defined by U.S. Army Medical Command (MEDCOM) policy 14-094; 18 Dec 2014).
* PTSD Checklist - Civilian (PCL-C) score of 32 or greater at screening
* Acceptable clinically indicated preoperative laboratory studies, per standard site-specific protocols

Exclusion Criteria:

* Prior Stellate Ganglion Block (SGB)
* Allergy to amide local anesthetics (e.g., ropivacaine, bupivacaine)
* Pregnancy (evaluated by urine test pre-procedure)
* Current anticoagulant use
* History of a bleeding disorder
* Infection or mass at injection site
* Myocardial infarction within 6 months of procedure
* Phrenic or laryngeal nerve palsy (hoarseness)
* History of glaucoma
* History of schizophrenia, other psychotic disorder, bipolar disorder, or personality disorder (axis 2)
* Moderate or severe traumatic brain injury
* Symptoms of moderate to severe substance use disorder in past 30 days
* Suicidal ideation in the past 2 months, documented by the M.I.N.I.-Plus Suicidality Items
* Any ongoing other major life stressor or condition not listed here that the site Investigator believes clearly would place the participant at risk for injury or a poor outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Tripler Army Medical Center (TAMC), Honolulu, Hawaii
  - Womack Army Medical Center (WAMC), Fort Bragg, North Carolina
- Landstuhl Regional Medical Center (LRMC), Landstuhl, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rae Olmsted KL, Bartoszek M, Mulvaney S, McLean B, Turabi A, Young R, Kim E, Vandermaas-Peeler R, Morgan JK, Constantinescu O, Kane S, Nguyen C, Hirsch S, Munoz B, Wallace D, Croxford J, Lynch JH, White R, Walters BB. Effect of Stellate Ganglion Block Treatment on Posttraumatic Stress Disorder Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):130-138. doi: 10.1001/jamapsychiatry.2019.3474. PMID 31693083
- [Derived] Blakey SM, Rae Olmsted KL, Hirsch S, Asman K, Wallace D, Olmsted MG, Vandermaas-Peeler R, Karg RS, Walters BB. Differential posttraumatic stress disorder symptom cluster response to stellate ganglion block: secondary analysis of a randomized controlled trial. Transl Psychiatry. 2024 May 29;14(1):223. doi: 10.1038/s41398-024-02926-8. PMID 38811568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 123 participants screened eligible and completed the baseline CAPS-5
Pre-assignment Details: 113 participants were randomized to treatment/sham and underwent the study procedure at Week 0 and Week 2.
Period: Overall Study
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Started | 74 | 39
Week 2 Visit | 74 | 39
Week 4 Visit | 73 | 38
Week 6 Visit | 73 | 38
Week 8 Visit | 71 | 38
Final CAPS | 70 | 38
Completed | 70 | 38
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment | Total
Number analyzed (Participants) | 74 | 39 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 39 | 113
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 64 | 36 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Marital Status [Count of Participants; unit: Participants]
  Married | 67 | 33 | 100
  Unmarried | 7 | 6 | 13
Military Rank [Count of Participants; unit: Participants]
  Junior Enlisted | 3 | 3 | 6
  Non-commissioned Officer | 27 | 11 | 38
  Senior Enlisted | 28 | 19 | 47
  Warrant Officer | 5 | 3 | 8
  Commissioned Officer | 11 | 3 | 14
Met CAPS-5 Criteria for PTSD [Count of Participants; unit: Participants] — The CAPS-5 is a 30-item structured interview, administered by a credentialed behavioral health practitioner, that corresponds to the DSM-5 criteria for PTSD (Weathers et al. 2013, The Clinician Administered PTSD Scale for DSM-5, Boston MA: The National Center for PTSD).
  Participants | 60 | 31 | 91

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Score (CAPS-5) TSSS
Description: ≥ 10 point mean Clinician-Administered PTSD Scale for DSM 5 (CAPS 5) total symptom severity scores (TSSS) improvement from baseline to 8 weeks, adjusted for site and baseline TSSS (planned a priori), following paired SGB at 0 and 2 weeks. On the CAPS 5, the range for TSSS is 0 to 80, with higher scores indicating worse PTSD symptomatology. The CAPS-5 is a 30-item structured interview, administered by a credentialed behavioral health practitioner, that corresponds to the DSM-5 criteria for PTSD (Weathers et al. 2013, The Clinician Administered PTSD Scale for DSM-5, Boston MA: The National Center for PTSD).
Time Frame: Baseline, 8-weeks
Population: Multiple imputation performed for missing data; Mean change - Adjusted for site and baseline CAPS TSSS; adjusted mean reduction in TSSS from baseline to week 8 by treatment group from per-protocol analysis and secondary analysis among those who fulfilled CAPS 5 diagnostic criteria for PTSD at baseline were consistent with those from ITT analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 37.61 (11.13) | 39.82 (14.23)
  8-week follow-up | 25.67 (14.13) | 33.68 (15.60)

2. Secondary Outcome: PTSD Checklist (PCL-5)
Description: to evaluate symptoms measured by PTSD Checklist (PCL-5) at baseline; On the PCL 5, the range is 0 to 80, with higher scores indicating worse PTSD symptomatology.
Time Frame: Baseline, 8-weeks
Population: Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 41.54 (14.03) | 43.23 (18.13)
  8-week follow-up | 29.49 (19.29) | 38.11 (18.23)

3. Secondary Outcome: PTSD Checklist Civilian (PCL-C)
Description: to evaluate symptoms measured by PTSD Checklist Civilian (PCL-C) at baseline; The total symptom severity score ranges from 17 to 85. The higher the score, the more severe the PTSD symptomatology
Time Frame: Baseline, 8-weeks
Population: Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 53.30 (13.64) | 54.95 (15.67)
  8-week follow-up | 42.41 (17.47) | 50.65 (17.04)

4. Secondary Outcome: Mini-International Neuropsychiatric Interview (M.I.N.I.-Plus) Suicidality Items
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by Mini-International Neuropsychiatric Interview (M.I.N.I.-Plus) Suicidality Items at 8 weeks. The higher the score, the more severe the pathology. If an individual answers "yes" to any of seven initial questions concerning suicidal ideation in the past two months, they are asked an additional four questions regarding current suicidal ideation. Any positive answer on these four current questions triggers an automated alert system.
Time Frame: Baseline, 8-weeks
Measure: Median (Full Range); unit: number of events
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
number of events
  Baseline | 0 [0 to 3] | 0 [0 to 3]
  8-week follow-up | 0 [0 to 3] | 0 [0 to 4]

5. Secondary Outcome: Alcohol Use Disorders Identification Test (AUDIT/AUDIT-C)
Description: to evaluate symptoms measured by the Alcohol Use Disorders Identification Test at 8 weeks. Based on a scale of 0 to 12, a score of 4 or greater is considered positive in males, while a score of 3 or more is positive among females.
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 2.74 (2.64) | 3.18 (4.26)
  8-week follow-up | 2.72 (2.71) | 2.62 (3.80)

6. Secondary Outcome: Kessler Psychiatric Distress Scale (K6)
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by the Kessler Psychiatric Distress Scale (K6) at 8 weeks. Scores range from 0 to 24 resulting from 6 items administered on a scale of 0 to 4, with a score of 13 or greater indicative of serious psychological distress in the U.S. general population.
Time Frame: Baseline, 8-weeks
Population: Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 10.08 (5.55) | 10.33 (6.01)
  8-week follow-up | 7.80 (6.41) | 10.00 (6.25)

7. Secondary Outcome: The Patient Health Questionnaire (PHQ-9)
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by The Patient Health Questionnaire (PHQ-9) at 8 weeks; On the PHQ-9, the range is 0 to 27, with higher scores indicating worse depression symptomatology.
Time Frame: Baseline, 8-weeks
Population: Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 12.57 (6.05) | 12.69 (6.61)
  8-week follow-up | 8.68 (6.02) | 11.76 (6.25)

8. Secondary Outcome: Generalized Anxiety Disorder 7-item Survey (GAD-7)
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by Generalized Anxiety Disorder 7-item survey (GAD-7) at 8 weeks;On the GAD-7, the range is 0 to 21, with higher scores indicating worse anxiety symptomatology.
Time Frame: Baseline, 8-weeks
Population: Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 12.39 (5.35) | 12.49 (5.50)
  8-week follow-up | 8.11 (6.02) | 11.19 (6.38)

9. Secondary Outcome: 12-item Short Form Survey (SF-12) of Physical Functioning
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by 12-item Short Form Survey (SF-12) at 8 weeks. The score mean is 50; standard deviation of 10. The physical component score (PCS-12) is one of two summary scores reported for the SF-12. Higher scores indicate better physical health. The United States population average PCS-12 is 50 points.
Time Frame: Baseline, 8-weeks
Population: Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 41.04 (8.16) | 42.01 (7.87)
  8-week follow-up | 43.43 (8.33) | 41.28 (8.18)

10. Secondary Outcome: Short Pain Scale
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by the Short Pain Scale at 8 weeks; On the pain rating, the range is 0 to 10, with higher scores indicating worse pain.
Time Frame: Baseline, 8-weeks
Population: [*] Analysis Population Description Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 4.61 (2.40) | 4.95 (2.21)
  8-week follow-up | 4.10 (2.51) | 4.86 (2.30)

11. Secondary Outcome: Current Medications
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by a decrease in Current Medications at 8 weeks; in order to assess the potential impact of medication use concurrent with study participation, information on prescription psychotropics (including stimulants, anxiolytics, and antidepressants), anticonvulsants, antipsychotics, anticholinergic drugs, opioids, nicotine, sleeping medications, antihypertensives, and sympathomimetics/sympatholytics was collected.
Time Frame: Baseline, 8-weeks
Measure: Median (Full Range); unit: Medications
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
Medications
  Baseline | 1 [0 to 12] | 2 [0 to 6]
  8-week follow-up | 1 [0 to 13] | 1 [0 to 5]

12. Secondary Outcome: 12 Item Short Form Survey (SF-12) of Mental Functioning
Description: to evaluate whether right-sided stellate ganglion block (SGB) performed at 0 and 2 weeks will result in improvement in symptoms measured by the Short Mental Functioning Scale at 8 weeks. The score mean is 50; standard deviation of 10. The mental component score (MCS-12) is one of two summary scores reported for the SF-12. Higher scores indicate better mental health. The United States population average MCS-12 is 50 points.
Time Frame: Baseline, 8-weeks
Population: Adjusted for site, gender, age, visit, and interaction between visit and treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
Number analyzed (Participants) | 74 | 39
score on a scale
  Baseline | 41.24 (11.32) | 40.16 (9.84)
  8-week follow-up | 42.83 (10.22) | 40.17 (9.50)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for eight weeks.
Arm/Group | Stellate Ganglion Block (SGB) | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/39
Other Adverse Events (participants affected / at risk) | 5/74 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stellate Ganglion Block (SGB) (N=74) | Sham Treatment (N=39)
Temporary irritation of larynx which resulted in coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain and redness at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vasovagal syncope with insertion of the IV (Nervous system disorders) | 1 (1) | 0 (0)
Detection of nodule or cyst (< 1 cm) in thyroid gland (Endocrine disorders) | 1 (1) | 0 (0)
Self-resolving episode of bradycardia (30-second duration; minimum heart rate of 32) (Cardiac disorders) | 1 (1) | 0 (0)
Report of mild, relative increase in pre-existing right tinnitus (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Treating physicians unblinded; Horner syndrome noticeable; specific population re psychotropic usage, administrative evaluations, TBI history; overall PTSD symptom severity low-moderate; a number of participants still fulfil PTSD criteria at 8 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03077919/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT03077919/SAP_001.pdf